CLINICAL TRIAL: NCT02489539
Title: Assessment of the GORE® EXCLUDER® Conformable AAA Endoprosthesis in the Treatment of Abdominal Aortic Aneurysms
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAA 13-03 (1); NCT02489552 (obsolete NCT alias)
Record Dates: First submitted 2015-06-22; First posted 2015-07-03 (Estimated); Results first posted 2024-04-04 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2024-12

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: Aortic aneurysm; Abdominal aorta; Stent graft; Aneurysm; Vascular Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aortic Aneurysm; Aneurysm; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Short Neck Substudy (Experimental): Subjects with abdominal aortic aneurysms having infrarenal aortic neck angulation ≤ 60˚ and infrarenal aortic neck length ≥10 mm treated with the GORE® EXCLUDER® Conformable AAA Endoprosthesis.
  Interventions: Device: GORE® EXCLUDER® Conformable AAA Endoprosthesis
- High Neck Angulation Substudy (Experimental): Subjects with abdominal aortic aneurysms having infrarenal aortic neck angulation > 60˚ and ≤ 90˚ and infrarenal aortic neck length ≥10 mm treated with the GORE® EXCLUDER® Conformable AAA Endoprosthesis.
  Interventions: Device: GORE® EXCLUDER® Conformable AAA Endoprosthesis

INTERVENTIONS:
Device: GORE® EXCLUDER® Conformable AAA Endoprosthesis — Endovascular Aneurysm repair (EVAR) is a minimally invasive procedure designed to exclude an aneurysmal segment of the aorta from blood circulation. The EVAR procedure involves delivery of a stent- graft compressed onto a catheter to an aneurysmal segment of the aorta from a remote access site, generally the femoral artery. Arterial access may be done by either percutaneous or cut-down technique.

SUMMARY:
The purpose of the study is to assess the safety and effectiveness of the GORE® EXCLUDER® Conformable AAA Endoprosthesis to treat an infrarenal aneurysm located in the abdominal aorta. Performance of the GORE® EXCLUDER® Conformable AAA Endoprosthesis will be judged by separate performance goals.

DETAILED DESCRIPTION:
The study design is a prospective, nonrandomized, international, multicenter study comprised of two parallel substudies. The total subject population is 175 subjects with 80 subjects assigned to the Short Neck Substudy and 95 subjects to the High Neck Angulation Substudy.

This clinical study will include up to fifty-six sites in the US. Each enrolled subject will undergo periodic follow-up evaluations involving physical exams and contrast-enhanced computed tomography (CT) scans at specific, protocol-defined intervals for a period of five years following the GORE® EXCLUDER® Conformable AAA Endoprosthesis implant. Each Substudy will be evaluated and reported independently from each other according to the Safety and Effectiveness Endpoints. No comparative analyses between these substudies are planned.

ELIGIBILITY:
Inclusion Criteria:

1. AAA meeting any of the following criteria:

   * Maximum diameter ≥50 mm
   * Rapid growth (>5 mm in a 6 month period)
   * Non-ruptured AAA presenting with clinical symptoms
2. Adequate anatomy to receive the GORE® EXCLUDER® Conformable AAA Endoprosthesis, including:

   * Adequate iliac / femoral access
   * Infrarenal aortic neck diameter 16-32 mm
   * Infrarenal aortic neck length ≥10 mm
   * Aortic neck angle ≤ 90˚
   * Distal iliac artery seal zone ≥10 mm
   * Iliac artery diameter 8-25 mm
3. An Informed Consent Form (ICF) signed by Subject
4. Male or infertile female
5. Able to comply with Protocol requirements including following-up
6. Life expectancy > 2 years
7. Age ≥ 21 years

Exclusion Criteria:

1. Mycotic or ruptured aneurysm
2. Known concomitant thoracic aortic aneurysm which requires surgical intervention
3. Renal insufficiency defined as creatinine > 2.5 mg/dL or patient undergoing dialysis
4. New York Heart Association (NYHA) class IV
5. Aneurysmal, dissected, heavily calcified, or heavily thrombosed landing zone(s)
6. Severely tortuous or stenotic iliac and / or femoral arteries
7. Patient has body habitus or other medical condition which prevents adequate delineation of the aorta
8. Participating in another investigational device or drug study within 1 year of treatment
9. Systemic infection which may increase the risk of endovascular graft infection
10. Known degenerative connective tissue disease, e.g., Marfan or Ehler-Danlos Syndrome
11. Planned concomitant surgical procedure or major surgery within 30 days of treatment date
12. Known history of drug abuse
13. Known sensitivities or allergies to the device materials

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2027-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Rhee, MD, Principal Investigator — Maimonides Medical Center (US)
Locations (51):
- United States (51):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - Leland Stanford Junior University, Stanford, California
  - River City Clinical Research, Jacksonville, Florida
  - Baptist Cardiac and Vascular Institute, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - Sarasota Vascular Specialists, Sarasota, Florida
  - Emory University, Atlanta, Georgia
  - Vascular Surgical Associates, PC, Marietta, Georgia
  - Loyola University - Chicago, Maywood, Illinois
  - Southern Illinois University, Springfield, Illinois
  - University of Iowa Hospitals & Clinic, Iowa City, Iowa
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Spectrum Health System, Grand Rapids, Michigan
  - Essentia Institute of Rural Health, Duluth, Minnesota
  - Minneapolis Heart Institute Foundation - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Minneapolis Radiology and Vascular Research Foundation, Plymouth, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine - St. Louis, St Louis, Missouri
  - Mercy Research, St Louis, Missouri
  - The Hitchcock Foundation, Lebanon, New Hampshire
  - AHA Hospital Corp., Morristown, New Jersey
  - Maimonides Medical Center, Brooklyn, New York
  - Research Foundation SUNY Buffalo, Buffalo, New York
  - Staten Island University Hospital, Staten Island, New York
  - Mission Hospital, Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Moses Cone Memorial Hospital, Greensboro, North Carolina
  - NC Heart and Vascular Research, LLC, Raleigh, North Carolina
  - Good Samaritan Hospital-Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Oklahoma Heart Hospital Research Foundation, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health-Upstate, Greenville, South Carolina
  - Sanford Clinic - Clinic Research, Sioux Falls, South Dakota
  - North Central Heart Institute, Ltd., Sioux Falls, South Dakota
  - University of Tennessee, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Heart Institute/Baylor St. Luke's Medical Center, Houston, Texas
  - The Methodist Hospital - Houston, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Sentara Medical Group, Norfolk, Virginia
  - Inova Cardiology-Fairfax, Virginia Beach, Virginia
  - CAMC Health Education and Research Institute, Inc., Charleston, West Virginia
  - University of Wisconsin System, Madison, Wisconsin
  - Aurora Health Care, Metro Inc., Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Device and aneurysm status will be communicated to subject through standard of care evaluations. Core Lab data will not be available to subjects.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Short Neck Substudy | High Neck Angulation Substudy
Started | 80 | 95
Completed | 78 | 0
Not Completed | 2 | 95

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Short Neck Substudy | High Neck Angulation Substudy | Total
Number analyzed (Participants) | 80 | 95 | 175
Age, Continuous [Median (Full Range); unit: years] | 73 [56 to 96] | 74 [59 to 92] | 74 [56 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 24 | 33
  Male | 71 | 71 | 142
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 75 | 87 | 162
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States | 80 | 95 | 175

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Free From Primary Safety Endpoint Event
Description: The primary safety endpoint event includes a composite of the following:
  * Death
  * Stroke
  * Myocardial Infarction
  * Bowel Ischemia
  * Paraplegia
  * Respiratory Failure
  * Renal Failure
  * Procedural Blood Loss > 1000 mL
  * Thromboembolic events (including limb occlusion and distal embolic events)
Time Frame: 30 Days
Population: This population consists of subjects with a physical exam follow-up visit at or after 30 days following CEXC device implant procedure. Additionally, any subjects with an eligible safety event, even if they did not complete a follow-up visit at or after 30 days following implant procedure, were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Short Neck Substudy | High Neck Angulation Substudy
Number analyzed (Participants) | 79 | 92
Participants | 79 | 89

2. Primary Outcome: Number of Subjects With Device Treatment Success
Description: The Primary Effectiveness Endpoint of device treatment success is a composite of technical success (successful access and deployment of all required GORE® EXCLUDER® Conformable AAA Endoprosthesis components) and freedom from:
  * Type I endoleak in the 12 month window
  * Type III endoleak in the 12 month window
  * Migration (10 mm or more) at the 12 month window (relative to post-operative baseline)
  * AAA enlargement ≥5 mm with or without intervention at the 12 month window (relative to post-operative baseline)
  * AAA rupture through the 12 month window
  * Conversion to open repair through the 12 month window
Time Frame: 12 Months
Population: This population consists of subjects with both a post-op contrast-enhanced CT (CTA) and a 12-Month CTA. Additionally, any subjects with an eligible effectiveness event, even if they did not complete the necessary follow-up visit or imaging to otherwise be included in the population, were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Short Neck Substudy | High Neck Angulation Substudy
Number analyzed (Participants) | 66 | 77
Participants | 65 | 73

3. Secondary Outcome: Number of Subjects With Reintervention
Description: Defined as an adverse event treatment performed to either treat the abdominal aneurysm and/or device-related complication (Adjudicated by independent Clinical Events Committee)
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

4. Secondary Outcome: Number of Subjects With Stent Fracture
Description: Defined as fracture of the wire used to construct the stent (assessed by independent 3rd party imaging laboratory)
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

5. Secondary Outcome: Number of Subjects With Type II Endoleak
Description: Defined as an endoleak arising from a patent branch vessel perfusing the aneurysm, e.g., lumbar or inferior mesenteric branch. (assessed by independent 3rd party imaging laboratory)
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

6. Secondary Outcome: Number of Subjects With Aneurysm-related Mortality
Description: Defined as a composite of the following: death within 30 days or in hospital from initial procedure, death due to rupture of the originally treated aneurysm and death within 30 days or in hospital following a procedure to treat the originally treated aneurysm. (Adjudicated by independent Clinical Events Committee)
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

7. Secondary Outcome: Number of Subjects With Significant Index Procedure Blood Loss
Description: Defined as estimated blood loss recorded during the endovascular procedure > 1000 mL
Time Frame: Procedure Day
Population: Subjects with non-missing procedural blood loss
Measure: Count of Participants; unit: Participants
Arm/Group | Short Neck Substudy | High Neck Angulation Substudy
Number analyzed (Participants) | 80 | 93
Participants | 0 | 3

8. Secondary Outcome: Number of Subjects With Type IV Endoleak
Description: Defined as Endoleak of whole blood through the graft fabric (Graft Porosity). (assessed by independent 3rd party imaging laboratory)
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

9. Secondary Outcome: Median Hospital Stay
Description: Defined as time to discharge for initial procedural hospitalization
Time Frame: Through initial hospital discharge
Population: All enrolled subjects
Measure: Median (Full Range); unit: days
Arm/Group | Short Neck Substudy | High Neck Angulation Substudy
Number analyzed (Participants) | 80 | 95
days | 1.0 [1 to 4] | 1.0 [1 to 13]

10. Secondary Outcome: Median Index Procedure Time
Description: Defined as time from first arterial access in the groin to the closure of the final access vessel
Time Frame: Procedure Day
Population: All enrolled subjects
Measure: Median (Full Range); unit: minutes
Arm/Group | Short Neck Substudy | High Neck Angulation Substudy
Number analyzed (Participants) | 80 | 95
minutes | 84.0 [33 to 251] | 110 [40 to 358]

11. Secondary Outcome: Number of Subjects With Severe Stroke
Description: Defined as stroke resulting in severe impairment or fatal outcome (Adjudicated by independent Clinical Events Committee)
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

12. Secondary Outcome: Number of Subjects With Severe Myocardial Infarction
Description: Defined as myocardial Infarction resulting in severe hemodynamic dysfunction necessitating resuscitation, cardiac arrest, or fatal outcome. (Adjudicated by independent Clinical Events Committee)
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

13. Secondary Outcome: Number of Subjects With Severe Bowel Ischemia
Description: Defined as bowel Ischemia resulting in bowel resection or fatal outcome (Adjudicated by independent Clinical Events Committee)
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

14. Secondary Outcome: Number of Subjects With Severe Paraplegia
Description: Paraplegia resulting in major permanent deficit (Adjudicated by independent Clinical Events Committee)
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

15. Secondary Outcome: Number of Subject Deaths
Description: Defined as death of any cause (all-cause mortality)
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

16. Secondary Outcome: Number of Subjects With Severe Renal Failure
Description: Defined as renal failure resulting in permanent dialysis, transplant, or fatal outcome (Adjudicated by independent Clinical Events Committee)
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

17. Secondary Outcome: Number of Subjects With Severe Respiratory Failure
Description: Defined as respiratory failure resulting in prolonged intubation (> 48 hours), tracheostomy, deterioration in pulmonary function, new onset O2 dependence, or fatal outcome (Adjudicated by independent Clinical Events Committee)
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

18. Secondary Outcome: Number of Subjects With Thromboembolic Events (Including Limb Occlusion and Distal Embolic Events)
Description: Defined as ischemic events from tissues distal to the device implantation site (lower extremity, buttock, etc.) and that are a direct result of an occlusion within the device or sufficiently debilitating to necessitate bypass, open surgical repair, or limb amputation (Adjudicated by independent Clinical Events Committee)
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

19. Secondary Outcome: Number of Subjects With Type I Endoleak
Description: Defined as endoleak arising from the proximal (Type IA) or distal (Type IB) sealing zone of the device perfusing the aneurysm. (assessed by independent 3rd party imaging laboratory)
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

20. Secondary Outcome: Number of Subjects With Type III Endoleak
Description: Defined as endoleak arising from the component junction(s) of the prosthesis or due to damage to the graft material (assessed by independent 3rd party imaging laboratory)
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

21. Secondary Outcome: Number of Subjects With Migration
Description: Defined as prosthesis and/or intercomponent migration (10 mm or more) relative to post-operative baseline (assessed by independent 3rd party imaging laboratory)
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

22. Secondary Outcome: Median Procedural Blood Loss (mL)
Description: Median blood loss at index procedure
Time Frame: Procedure Day
Population: Number of subjects with non-missing blood loss
Measure: Median (Full Range); unit: mL
Arm/Group | Short Neck Substudy | High Neck Angulation Substudy
Number analyzed (Participants) | 80 | 93
mL | 50 [0 to 1000] | 50 [0 to 2700]

23. Secondary Outcome: Number of Subjects With AAA Enlargement ≥5 mm
Description: Defined as AAA enlargement ≥5 mm (with or without reintervention) relative to post-operative baseline (assessed by independent 3rd party imaging laboratory)
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

24. Secondary Outcome: Number of Subjects With Abdominal Aortic Aneurysm Rupture
Description: Defined as rupture in the treated segment of the aorta verified with direct observation or CT scan
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

25. Secondary Outcome: Number of Subjects With Conversion to Open Repair
Description: Defined as open surgical abdominal aneurysm repair necessitating the explant of the stent-graft and abdominal aortic reconstruction (Adjudicated by independent Clinical Events Committee)
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-12

26. Secondary Outcome: Technical Success
Description: Successful access and deployment of all required CEXC device components, comprised of all the following:
  * Successful access
  * Successful deployment of Device endoprostheses in the intended anatomical location
  * Successful removal of all device delivery catheters from the patient
  * Patent Device components on completion angiography
  * Absence of Type I or Type III endoleak on completion angiography
  * Successful access site closure
Time Frame: Procedure Day
Population: All enrolled subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Short Neck Substudy | High Neck Angulation Substudy
Number analyzed (Participants) | 80 | 95
Participants | 80 | 93

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Short Neck Substudy | High Neck Angulation Substudy
All-Cause Mortality (participants affected / at risk) | 15/80 | 25/95
Serious Adverse Events (participants affected / at risk) | 48/80 | 57/95
Other Adverse Events (participants affected / at risk) | 32/80 | 48/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Short Neck Substudy (N=80) | High Neck Angulation Substudy (N=95)
Acute anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 6 (6)
Symptomatic anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute decompensated heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2)
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure aggravated (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Chronic diastolic heart failure (Cardiac disorders) | 0 (0) | 1 (2)
Chronic heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Congestive cardiac failure aggravated (Cardiac disorders) | 0 (0) | 3 (3)
Congestive heart failure (Cardiac disorders) | 1 (1) | 2 (2)
Coronary artery disease (Cardiac disorders) | 2 (2) | 1 (1)
Coronary artery disease aggravated (Cardiac disorders) | 1 (1) | 0 (0)
Heart attack (Cardiac disorders) | 0 (0) | 1 (1)
Heart block third degree (Cardiac disorders) | 1 (1) | 0 (0)
Junctional bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Left anterior fascicular block (Cardiac disorders) | 0 (0) | 1 (1)
Mitral regurgitation (Cardiac disorders) | 0 (0) | 1 (1)
Non ST segment elevation myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Non STEMI (Cardiac disorders) | 1 (1) | 0 (0)
Non-sustained ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Persistent atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Right bundle branch block (Cardiac disorders) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Acute diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colovesical fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Distress gastrointestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal bleeding (Gastrointestinal disorders) | 2 (2) | 0 (0)
Mouth bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancreatitis acute on chronic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small bowel obstruction (Gastrointestinal disorders) | 2 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Edema of lower extremities (General disorders) | 1 (1) | 0 (0)
Endotension (General disorders) | 1 (1) | 0 (0)
General debility (General disorders) | 1 (1) | 0 (0)
Incarcerated hernia (General disorders) | 0 (0) | 1 (1)
Stent-graft endoleak type IA (General disorders) | 1 (1) | 0 (0)
Stent-graft endoleak type IB (General disorders) | 0 (0) | 2 (2)
Stent-graft endoleak type II (General disorders) | 2 (2) | 4 (5)
Unknown cause of death (General disorders) | 2 (2) | 4 (4)
Weakness generalized (General disorders) | 3 (3) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Mirizzi syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1)
Aspiration pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bloodstream infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis of leg (Infections and infestations) | 0 (0) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Community acquired pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Influenza A virus infection (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 5 (7)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Recurrent urinary tract infection (Infections and infestations) | 1 (2) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Septic pulmonary embolism (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 4 (4) | 2 (2)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Femoral artery pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fractured ribs (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site ecchymosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury to iliac artery (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar spine compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative delirium (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative fever (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic spine compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture T9 (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic hemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Elevated prostate specific antigen [PSA] (Investigations) | 1 (1) | 0 (0)
Fibrin D dimer increased (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Chest wall hematoma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Degenerative joint disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hip arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hips osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Appendix cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon adenomatous polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Endometrial carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Liver metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Lung metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm of descending colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic gastric adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic neoplasm of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm urinary bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Progression of prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Spinal metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Unknown primary cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Alzheimer's disease (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (2)
Internal carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Lightheadedness (Nervous system disorders) | 1 (1) | 0 (0)
Memory loss (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Middle cerebral artery stroke (Nervous system disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 3 (3)
Transient ischemic attack (Nervous system disorders) | 1 (2) | 2 (2)
VIth nerve palsy (Nervous system disorders) | 0 (0) | 1 (2)
Device kink (Product Issues) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 3 (3)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute renal insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic renal insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1)
End stage renal disease (ESRD) (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Impaired renal function (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery dissection (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery occlusion (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5)
Acute on chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Exacerbation of asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Unilateral pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Venous stasis ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pacemaker battery replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Arterial bleeding (Vascular disorders) | 0 (0) | 1 (1)
Arterial stenosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis leg (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Lower limb ischemia (Vascular disorders) | 0 (0) | 1 (1)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Popliteal artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Popliteal artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Refractory shock (Vascular disorders) | 1 (1) | 0 (0)
Type A aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Short Neck Substudy (N=80) | High Neck Angulation Substudy (N=95)
Stent-graft endoleak type II (General disorders) | 32 (38) | 44 (46)
Urinary tract infection (Infections and infestations) | 2 (2) | 8 (8)
Urinary retention (Renal and urinary disorders) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI(s) are restricted publishing multi-site aggregate trial results until the multi-center manuscript is published (Gore reserves the right to extend (as applicable) if filing a patent application). Prior to publication, Gore is allowed 60 day review period and the right to remove proprietary information.

DOCUMENTS (2):
  • Study Protocol (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/39/NCT02489539/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/39/NCT02489539/SAP_001.pdf